CLINICAL TRIAL: NCT05327101
Title: Quantifying Patient Preferences for Leadless Pacemaker Devices
Brief Title: Patient Preferences for Leadless Pacemakers
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10435
Record Dates: First submitted 2022-04-04; First posted 2022-04-14 (Actual); Results first posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Rhythm Disorder; Bradycardia; Cardiac Pacemaker Artificial
MeSH Terms: conditions — Arrhythmias, Cardiac; Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Other: Patient Preference Survey — Patient preference survey on implantable cardiac pacemaker systems

SUMMARY:
Prospective, non-randomized, multi-center study designed to quantify patient preferences pertaining to risks and features of conventional transvenous pacemakers and leadless pacemakers

DETAILED DESCRIPTION:
The purpose of this study is to quantify patient preferences pertaining to risks and features of conventional transvenous pacemakers and leadless pacemakers. The preference study is designed to elicit patient preferences for risks and features that vary between a dual chamber leadless pacemaker system and a dual chamber transvenous pacemaker system, to quantify their relative importance.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and speak English to consent to participate in the survey
* Willing and able to use a tablet or computer to complete the survey
* Scheduled to undergo evaluation for a de novo cardiac pacemaker at the study site (patient may or may not have a known indication for a pacemaker at the time)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 300 patients
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shelby Reed, PhD, Principal Investigator — Duke Clinical Research Institute
Locations (11):
- United States (11):
  - Honor Health, Scottsdale, Arizona
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Pacific Heart Institute, Santa Monica, California
  - Baptist Medical Center, Jacksonville, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Prairie Education & Research Cooperative, Springfield, Illinois
  - Charlton Memorial Hospital, Fall River, Massachusetts
  - New York Presbyterian Hospital/Cornell University, New York, New York
  - Hightower Clinical, Oklahoma City, Oklahoma
  - University of Utah Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Reed SD, Yang JC, Wallace MJ, Sutphin J, Johnson FR, Ozdemir S, Delgado SM, Goates S, Harbert N, Lo M, Rajagopalan B, Ip JE, Al-Khatib SM. Patient Preferences for Features Associated With Leadless Versus Conventional Transvenous Cardiac Pacemakers. Circ Cardiovasc Qual Outcomes. 2024 Dec;17(12):e011168. doi: 10.1161/CIRCOUTCOMES.124.011168. Epub 2024 Nov 21. PMID 39569505

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from Aveir™ DR IDE trial study sites. One-hundred seventeen patients were recruited and completed the survey instrument.
Groups:
- Patient Preferences Survey: Patients were recruited from Aveir™ DR IDE trial study sites. To minimize selection bias, patients meeting the criteria listed above and agreeing to participate were asked to complete the patient-preference survey before being approached about their potential interest in enrolling in the IDE trial. Thus, they completed the patient-preference survey before they received information about dual-chamber pacemakers from the site physician and/or the Aveir™ DR IDE study and before they received a pacemaker if they ultimately received one.
Period: Overall Study
Arm/Group | Patient Preferences Survey
Started | 117
Completed | 117
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Patient Preferences Survey: Patients were recruited from Aveir™ DR IDE trial study sites. To minimize selection bias, patients meeting specified criteria and agreeing to participate were asked to complete the patient-preference survey before being approached about their potential interest in enrolling in the IDE trial. Thus, they completed the patient-preference survey before they received information about dual-chamber pacemakers from the site physician and/or the Aveir™ DR IDE study and before they received a pacemaker if they ultimately received one.
Arm/Group | Patient Preferences Survey
Number analyzed (Participants) | 117
Age, Customized [Mean (Standard Deviation); unit: years] | 67.3 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 113
  Unknown or Not Reported | 2
Marital Status [Count of Participants; unit: Participants]
  Single/never married | 7
  Married/living as married | 81
  Divorced or separated | 19
  Widowed/surviving partner | 9
  Other | 1
Health Insurance [Number; unit: participants]
  Through a state or federal insurance exchange | 11
  Through my (or another person's) employer or union | 26
  Medicare alone | 27
  Medicare and supplemental insurance | 53
  Medicaid | 7
  Veterans affairs | 6
  Other | 1
  I do not have health insurance | 2
Highest Level of Education [Count of Participants; unit: Participants]
  Less than high school | 4
  Some high school | 3
  High school or equivalent (such as GED) | 19
  Some college but no degree | 22
  Technical school | 7
  Associate's degree or 2-year college degree | 16
  4-year college degree (such as BA, BS) | 26
  Some graduate school but no degree | 3
  Graduate or professional degree (such as MBA, MS, MA, MD, PhD) | 15
  Missing | 2
Height [Mean (Standard Deviation); unit: inches] | 67.8 (4.5)
Weight [Mean (Standard Deviation); unit: pounds] | 184.9 (43.5)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.1 (5.6)
Employment [Count of Participants; unit: Participants] — Count of participants selecting employment option. Participants allowed to select more than 1 option
  Participants
    Employed with hourly pay | 13
    Employed with salary | 18
    Self-employed | 9
    Homemaker | 4
    Student | 1
    Disabled | 11
    Not working but looking for a job | 1
    Not working and NOT looking for a job | 1
    Unable to work or on disability | 1
    Volunteer work | 3
    Other | 0
    Retired | 68
Race [Count of Participants; unit: Participants] — Count of participants selecting race option. Participants were allowed to select more than 1 option
  Participants
    American Indian or Alaska Native | 1
    Asian | 3
    Black or African American | 4
    Native Hawaiian or Other Pacific Islander | 0
    White | 110
    Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Rankings for Pacemaker Device Features
Description: Ranking of six pacemaker device features from most concerning (1) to least concerning (6)
Time Frame: Baseline
Population: Each respondent was asked to rank the six features (insertion procedure, pacemaker type, pacemaker location, no heavy lifting, scar on chest, and lump on chest) from most concerning (1) to least concerning (6). The table reports the mean ranking for each device feature evaluated on a scale from 1-6. The number of respondents is 90 because 27 respondents skipped the ranking questions
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Preferences Survey
Number analyzed (Participants) | 90
score on a scale
  Insertion procedure | 2.3 (1.3)
  Pacemaker type | 2.6 (1.2)
  Pacemaker location | 2.2 (1.0)
  No heavy lifting for 6 weeks | 4.7 (1.5)
  Scar on chest | 5.1 (1.0)
  Lump on chest | 4.1 (1.4)

2. Primary Outcome: Results From RPL Model of Discrete Choice Experiment Choice Questions - Preference Weights (Effect-coded Parameters)
Description: The preference weights for the RPL model. Effect-coded parameters generate log-odds preference weights representing the relative strength of preference for each attribute level versus the mean effect across levels normalized at zero. A higher weight indicates a more preferred level while a lower weight indicates a less preferred level.
Time Frame: Baseline
Measure: Number; unit: preference weights
Arm/Group | Patient Preferences Survey
Number analyzed (Participants) | 117
preference weights
  Pacemaker type - Leadless, removable | 0.340
  Pacemaker type - Leadless, non-removable | -0.310
  Pacemaker type - Transvenous | -0.030
  Battery life - 15 years | 0.454
  Battery life - 12 years | 0.253
  Battery life - 8 years | -0.235
  Battery life - 5 years | -0.473
  Time since regulatory approval - 10 years | 0.212
  Time since regulatory approval - 2 years | -0.212
  Discomfort for 6 months - No discomfort | 0.099
  Discomfort for 6 months - Discomfort | -0.099
  Risk of Complication - 1% | 0.957
  Risk of Complication - 5% | 0.396
  Risk of Complication - 10% | -0.390
  Risk of Complication - 20% | -0.963
  Risk of infection - 1% | 0.961
  Risk of infection - 5% | 0.408
  Risk of infection - 10% | -0.132
  Risk of infection - 20% | -1.237

3. Primary Outcome: Results From RPL Model of Discrete Choice Experiment Choice Questions- Standard Deviations
Description: The standard deviations representing the degree of variation in preference weights, with larger estimates representing preference heterogeneity.
Time Frame: Baseline
Measure: Number; unit: standard deviation
Arm/Group | Patient Preferences Survey
Number analyzed (Participants) | 117
standard deviation
  Pacemaker type - Leadless, removable | 0.490
  Pacemaker type - Leadless, non-removable | 1.411
  Pacemaker type - Transvenous | 0.921
  Battery life - 15 years | 0.562
  Battery life - 12 years | 0.420
  Battery life - 8 years | 0.242
  Battery life - 5 years | 0.741
  Time since regulatory approval - 10 years | 0.345
  Time since regulatory approval - 2 years | 0.345
  Discomfort for 6 months - No discomfort | 0.121
  Discomfort for 6 months - Discomfort | 0.121
  Risk of Complication - 1% | 0.606
  Risk of Complication - 5% | 0.346
  Risk of Complication - 10% | 0.838
  Risk of Complication - 20% | 1.790
  Risk of infection - 1% | 0.683
  Risk of infection - 5% | 0.293
  Risk of infection - 10% | 0.077
  Risk of infection - 20% | 1.052

4. Primary Outcome: Maximum-acceptable Risks of a Complication
Description: Maximum-acceptable risk (MAR) of a complication was calculated for patients based off latent-class analysis with two groups-leadless class and transvenous class (see secondary outcome Constrained 2-class Latent-class model preference weights). The MAR represents risk level patients would be willing to accept to obtain their preferred pacemaker type, no discomfort, a device with longer battery life, and a device with more time since regulatory approval.
Time Frame: Baseline
Measure: Number (95% Confidence Interval); unit: percentage of maximum-acceptable risk
Arm/Group | Patient Preferences Survey
Number analyzed (Participants) | 117
percentage of maximum-acceptable risk
  Patients in leadless class willing to accept MAR for removable leadless rather than transvenous | 13.4 [6.4 to 23.8]
  Patients in transvenous class willing to accept MAR for removable leadless rather than transvenous | 0 [0 to 0]
  Patients in leadless class willing to accept MAR for transvenous rather than removable leadless | 0 [0 to 0]
  Patients in transvenous class willing to accept MAR for transvenous rather than removable leadless | 7.6 [1.7 to 16.8]
  Patients in leadless class willing to accept MAR for transvenous rather than nonremovable leadless | 0 [0 to 0]
  Patients in transvenous class willing to accept MAR for transvenous instead of nonremovable leadless | 14.5 [7.3 to 36.6]
  Patients in leadless class willing to accept MAR for removable rather than nonremovable leadless | 5.1 [0.4 to 9.2]
  Patients in transvenous class willing to accept MAR for removable rather than nonremovable leadless | 6.3 [2.4 to 10.5]
  Transvenous class patients willing to accept MAR for 10 yrs since government approval rather than 2 | 0.7 [-2 to 3.7]
  Leadless class patients willing to accept MAR for 10 yrs since government approval rather than 2 | 6.8 [3.6 to 10.1]
  Leadless & transvenous class patients willing to accept MAR for 15 yrs of battery life instead of 2 | 6.7 [3.9 to 9.9]
  Leadless & transvenous class patients willing to accept MAR for no discomfort rather than discomfort | 2.0 [0.5 to 4.1]

5. Primary Outcome: Maximum-acceptable Risks of an Infection
Description: Maximum-acceptable risk (MAR) of an infection was calculated for patients based off latent-class analysis with two groups-leadless class and transvenous class (see secondary outcome Constrained 2-class Latent-class model preference weights). The MAR represent the risk that patients would be willing to accept to obtain their preferred pacemaker type, no discomfort, a device with longer battery life, and a device with more time since regulatory approval.
Time Frame: Baseline
Measure: Number (95% Confidence Interval); unit: percentage of maximum-acceptable risk
Arm/Group | Patient Preferences Survey
Number analyzed (Participants) | 117
percentage of maximum-acceptable risk
  Patients in leadless class willing to accept MAR for removable leadless rather than transvenous | 16.8 [7.6 to 28.9]
  Patients in transvenous class willing to accept MAR for removable leadless rather than transvenous | 0 [0 to 0]
  Patients in leadless class willing to accept MAR for transvenous rather than removable leadless | 0 [0 to 0]
  Patients in transvenous class willing to accept MAR for transvenous rather than removable leadless | 8.9 [1.5 to 21.6]
  Patients in leadless class willing to accept MAR for transvenous rather than nonremovable leadless | 0 [0 to 0]
  Patients in transvenous class willing to accept MAR for transvenous instead of nonremovable leadless | 17.8 [8.5 to 38.3]
  Patients in leadless class willing to accept MAR for removable rather than nonremovable leadless | 4.7 [0.5 to 11.5]
  Patients in transvenous class willing to accept MAR for removable rather than nonremovable leadless | 6.6 [2.4 to 13.3]
  Transvenous class patients willing to accept MAR for 10 yrs since government approval rather than 2 | 0.8 [-1.6 to 3.1]
  Leadless class patients willing to accept MAR for 10 yrs since government approval rather than 2 | 7.6 [3.5 to 14]
  Leadless & transvenous class patients willing to accept MAR for 15 yrs of battery life instead of 2 | 7.5 [3.8 to 12.6]
  Leadless & transvenous class patients willing to accept MAR for no discomfort rather than discomfort | 1.9 [0.6 to 3.6]

6. Primary Outcome: Probability of Choosing Specified Pacemakers - All 3 Profiles
Description: Preference weight estimates were used to calculate the predicted probabilities that patients would choose a hypothetical pacemaker profile out of three different pacemaker types- leadless pacemaker removable, leadless pacemaker non-removable, or pacemaker with leads. Attributes for each pacemaker profile were defined using historical or published values. Preference weights from the latent class model were used to compute the probability that respondents within each class preference would choose a pacemaker profile over another.
Time Frame: Baseline
Measure: Number (95% Confidence Interval); unit: percentage of probability
Arm/Group | Patient Preferences Survey
Number analyzed (Participants) | 117
percentage of probability
  Probability leadless class to choose profile: leadless pacemaker removable | 41.7 [31.2 to 50.5]
  Probability transvenous class to choose profile: leadless pacemaker removable | 8.0 [2.9 to 19.4]
  Probability leadless class to choose profile: leadless pacemaker non-removable | 27.4 [16.7 to 39.8]
  Probability transvenous class to choose profile: leadless pacemaker non-removable | 4.5 [1.7 to 10.9]
  Probability leadless class to choose profile: pacemaker with leads | 30.9 [16.9 to 48.9]
  Probability transvenous class to choose profile: pacemaker with leads | 87.5 [70.1 to 95.3]

7. Primary Outcome: Probability of Choosing Specified Pacemakers - Leadless Pacemaker Removable vs. Leadless Pacemaker Non-removable
Description: Preference weight estimates were used to calculate the predicted probabilities that patients would choose a hypothetical pacemaker profile out of three different pacemaker types- leadless pacemaker removable or leadless pacemaker non-removable. Attributes for each pacemaker profile were defined using historical or published values. Preference weights from the latent class model were used to compute the probability that respondents within each class preference would choose a pacemaker profile over another.
Time Frame: Baseline
Measure: Number (95% Confidence Interval); unit: percentage of probability
Arm/Group | Patient Preferences Survey
Number analyzed (Participants) | 117
percentage of probability
  Probability leadless class to choose profile: leadless pacemaker removable | 60.4 [48.7 to 70.7]
  Probability transvenous class to choose profile: leadless pacemaker removable | 64.0 [54.3 to 72.7]
  Probability leadless class to choose profile: leadless pacemaker non-removable | 39.6 [29.3 to 51.3]
  Probability transvenous class to choose profile: leadless pacemaker non-removable | 36 [27.3 to 45.7]

8. Primary Outcome: Probability of Choosing Specified Pacemakers - Leadless Pacemaker Removable vs. Pacemaker With Leads
Description: Preference weight estimates were used to calculate the predicted probabilities that patients would choose a hypothetical pacemaker profile out of three different pacemaker types- leadless pacemaker removable or pacemaker with leads. Attributes for each pacemaker profile were defined using historical or published values. Preference weights from the latent class model were used to compute the probability that respondents within each class preference would choose a pacemaker profile over another.
Time Frame: Baseline
Measure: Number (95% Confidence Interval); unit: percentage of probability
Arm/Group | Patient Preferences Survey
Number analyzed (Participants) | 117
percentage of probability
  Probability leadless class to choose profile: leadless pacemaker removable | 57.4 [39.6 to 73.7]
  Probability transvenous class to choose profile: leadless pacemaker removable | 8.4 [3 to 21.6]
  Probability leadless class to choose profile: pacemaker with leads | 42.6 [26.3 to 60.4]
  Probability transvenous class to choose profile: pacemaker with leads | 91.6 [78.3 to 97]

9. Primary Outcome: Probability of Choosing Specified Pacemakers - Leadless Pacemaker Non-removable vs. Pacemaker With Leads
Description: Preference weight estimates were used to calculate the predicted probabilities that patients would choose a hypothetical pacemaker profile out of three different pacemaker types- leadless pacemaker non-removable or pacemaker with leads. Attributes for each pacemaker profile were defined using historical or published values. Preference weights from the latent class model were used to compute the probability that respondents within each class preference would choose a pacemaker profile over another.
Time Frame: Baseline
Measure: Number (95% Confidence Interval); unit: percentage of probability
Arm/Group | Patient Preferences Survey
Number analyzed (Participants) | 117
percentage of probability
  Probability leadless class to choose profile: leadless pacemaker non-removable | 46.9 [26.2 to 69.1]
  Probability transvenous class to choose profile: leadless pacemaker non-removable | 4.9 [1.7 to 13.4]
  Probability leadless class to choose profile: pacemaker with leads | 53.1 [30.8 to 73.8]
  Probability transvenous class to choose profile: pacemaker with leads | 95.1 [86.6 to 98.2]

10. Secondary Outcome: Constrained 2-class Latent-class Model Preference Weights
Description: Latent-class (LC) analysis was used to identify systematically different preference patterns across respondents. LC analysis provides a unique set of estimates of preference weights for a prespecified number of preference classes. Respondents are probabilistically assigned to classes based on the similarity of their responses to the overall preference pattern identified in each class.
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Patient Preferences Survey
Number analyzed (Participants) | 117
percentage of participants
  Leadless Class | 50.5
  Transvenous class | 49.6

11. Secondary Outcome: Number of Discrete Choice Experiment Questions Answered
Description: Number of Discrete choice experiment (DCE) questions answered by 117 respondents who answered at least the first 8 DCE questions. After respondents answered 8 DCE questions, they were asked if they would like to complete 4 additional questions.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Preferences Survey
Number analyzed (Participants) | 117
Participants
  8 questions | 41
  12 questions | 76

12. Secondary Outcome: Association of Patient Characteristics With Membership in the Transvenous Class Versus the Leadless Class
Description: Respondent characteristics can be associated with class membership probabilities to "profile" the classes. These results show if respondents with certain characteristics are more likely to be in one class versus the other. The odds ratios of being in the transvenous class versus the leadless class for patient characteristics. Odds ratios greater than 1 indicate a higher likelihood of being in the class preferring transvenous pacemakers and pacemakers with longer time since government approval.
Time Frame: Baseline
Measure: Number; unit: odds ratio
Arm/Group | Patient Preferences Survey
Number analyzed (Participants) | 117
odds ratio
  Male | 1.15
  Age, per 1-year increase | 0.99
  BMI, per unit increase | 1.05
  Major surgery requiring hospitalization in the last 5 years | 1.55
  Sedentary lifestyle with light activity | 2.73
  Interaction of lifestyle and BMI | 0.98

ADVERSE EVENTS:
Time Frame: Serious and other [non-serious] adverse events were not collected or assessed as part of the study
Description: Serious and other [non-serious] adverse events were not collected or assessed as part of the study
Arm/Group | Patient Preferences Survey
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT05327101/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT05327101/SAP_001.pdf